CLINICAL TRIAL: NCT06389084
Title: Parents Together: Supporting Parents to Promote Healthy Behaviours in Children
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Catherine Birken, Senior Scientist, Staff Pediatrician, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 179939
Record Dates: First submitted 2024-04-24; First posted 2024-04-29 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Child Eating Behaviours; Child Nutrition; Early Child Development; Parenting
Keywords: child eating behaviours; child nutrition; parenting; early child development

STUDY DESIGN:
Intervention Model Description: Randomized control trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention/treatment (Experimental): One or two caregivers of each enrolled child will attend an 8-week virtual parent/caregiver education program delivered by a Public Health Nurse. Additionally, the Public Health Nurse will deliver up to 4 individual coaching calls designed to address participant-identified goals related to the group content. The coaching calls will focus on helping to apply the messages and skills from the group sessions and making community connections.
  Interventions: Behavioral: Parents Together parenting course
- Control (No Intervention): Participants randomized to the control group receive regular health care.

INTERVENTIONS:
Behavioral: Parents Together parenting course — parenting course and coaching calls
  Arms: Intervention/treatment

SUMMARY:
The Parents Together trial aims to determine if the Parents Together program consisting of virtual parent group sessions and coaching calls, will result in better health outcomes for children. The program which is facilitated by a Public Health Nurse seeks to encourage healthy lifestyle behaviours, help build strong family relationships, and promote child development and mental health.

DETAILED DESCRIPTION:
This study will determine whether an intervention combining group-based parenting skills training and public health nurse coaching calls with a focus on healthy eating behaviours and nutrition, activity and sleep, compared to regular health care will lead to improved eating behaviours, movement behaviours, health and mental health in children aged 2-5 years and their caregivers.

Healthy children will be identified through primary care practices participating in The Applied Reearch Group for Kids (TARGet Kids!). Families who participate in this study will be randomly assigned to one of the two study groups that will run for 6-months:

Group A: Receive 8 weeks of group parenting education sessions and up to 4 public health nurse coaching calls. Group B: Receive regular health care.

ELIGIBILITY:
Inclusion Criteria:

Child enrolled in the The Applied Reearch Group for Kids (TARGet Kids!) cohort study Family is able to participate in English

Exclusion Criteria:

Children with a sibling already enrolled in the study Children with severe developmental delay or disability

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 128 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Child eating behaviours | 6 months post-randomization
  Child Eating Behaviour Questionnaire (CEBQ)

SECONDARY OUTCOMES:
Dietary intake and food environment | 6 months post-randomization
  Parent reported measures of dietary intake, and food environment (based on the Canadian Community Health Survey)
Nutritional risk | 6 months post-randomization
  Nutrition Screeening Tool for Every Preschooler (NutriSTEP)
Physical Activity, Sedentary Time, Sleep Duration | 6 months post-randomization
  Parent reported measures of physical activity, sedentary time, and sleep duration (based on the Canadian Community Health Survey)
Physical activity | 6 months post-randomization
  Parent reported measures of physical activity, sedentary time, and sleep duration (based on the Canadian Community Health Survey)
Social and emotional development | 6 months post-randomization
  Strengths and Difficulty Questionnaire (SDQ)
Child development | 6 months post-randomization
  Ages and Stages Questionnaire-3 (ASQ-3)
Family psychosocial health | 6 months post-randomization
  Parenting Stress Index (PSI) and Patient Health Questionnaire (PHQ-9)
Parenting | 6 months post-randomization
  Parenting Scale
Parenting sense of competence | 6 months post-randomization
  Parenting Sense of Competency Scale-Revised (PSOC-R
sociodemographic, maternal and child characteristics | 6 months post-randomization
  parent self-reported income, maternal education, ethnicity, immigration status, and marital status, questions about parents health, exposures during pregnancy, family medical history (based on the Canadian Community Health Survey)
zBMI | 6 months post-randomization
  Measure the difference in age and sex-standardized BMI z-score (zBMI) using child height and weight
Waist circumference | 6 months post-randomization
  Measure waist circumference using a tape measure
Blood pressure | 6 months post-randomization
  Measurement of diastolic and systolic blood pressure in children
  Measurement of diastolic and systolic blood pressure in children
  Measurement of diastolic and systolic blood pressure in children
  Measurement of diastolic and systolic blood pressure in children

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Birken, MD, MSc, Principal Investigator — The Hospital for Sick Children
Locations (2):
- Canada (2):
  - St. Michaels Hospital Pediatric Outpatient Clinic, Toronto, Ontario
  - The Hospital for Sick Children, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No